CLINICAL TRIAL: NCT04463225
Title: Patterns of Alcohol Use and Suicide-related Thoughts Among Recently Discharged Veterans: Risk Factors Associated With the Military-to-Veteran Transition
Brief Title: The Network Study: Soldiers Connecting for Work and Health
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cornell University (Other)
Collaborators: University of Washington (Other); University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB0009650; W81XWH1920001;CDMRP-BA160401 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2020-06-24; First posted 2020-07-09 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Alcohol Use Disorder; Depression
Keywords: Negative Emotional States; Anxiety; Alcohol norms; Trauma; PTSD; Stress; Self-medication
MeSH Terms: conditions — Alcoholism; Depression; Anxiety Disorders; Wounds and Injuries; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: One group will receive three opportunities to engage with a personalized internet-delivered brief intervention over the course of seven months and the second group will not be granted access.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention condition (Other): Participants assigned to the intervention condition will be invited to engage with an internet-based intervention three times during the course of the study.
  Interventions: Other: Internet-Delivered Brief Intervention
- Control (No Intervention): The control group will not be offered the internet-based intervention.

INTERVENTIONS:
Other: Internet-Delivered Brief Intervention — The internet-delivered brief intervention developed for the study can be accessed via computers and mobile devices.. The intervention will employ assessment data to give study participants feedback on their drinking behavior and offer strategies to avoid risky behavior.
  Arms: Intervention condition

SUMMARY:
This study will examine the efficacy of an internet-based brief intervention designed to reduce risky behavior in Soldiers as they transition from Active Duty into the civilian workforce as a Veteran. Up to 700 soldiers intending to separate from the Army will be recruited, with the intention of drawing a final sample of 450 participants. Study participants will be randomly assigned to either the intervention or the control group, stratified by age and gender.

DETAILED DESCRIPTION:
The combination of alcohol use and negative emotional states is a particularly toxic combination for suicide risk. The current study examines changes in alcohol/drug use/misuse and depression as soldiers undergo the transition from Active Duty to Veteran and offers a personalized internet-based brief intervention intended to prevent/reduce alcohol misuse and depression in this population.

The study's objectives are to empirically quantify the form of changes that occur with respect to alcohol use and depression over the transition; to identify stable individual risk factors (e.g., personality, military experiences) and dynamic risk factors (e.g., changes in stressors and normative contexts over time) that may be associated with differential temporal patterns of suicide-related behavior (i.e., alcohol use/misuse) and cognition (i.e., depression); and lastly, to determine whether a simple, internet-delivered brief intervention shown can reduce risky behavior in the transitioning Veteran population.

ELIGIBILITY:
Inclusion Criteria:

* Is US solider intending to separate from active duty during the study enrollment period
* Intends to seek civilian employment
* Plans to live in US

Exclusion Criteria:

* Plans to retire and not seek civilian employment
* Plans to live outside of the US
* Is separating or retiring from the National Guard or Reserves

Ages: 18 Years to 62 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The study will recruit up to 700 soldiers intending to separate from the Army in the initial phase of the study with the intention of securing a final sample of 450. Of the 450, 400 will be selected regardless of gender, but an additional 50 female soldiers will be recruited intentionally.
Enrollment: 450 (Estimated)
Dates: Start 2021-03-30 (Actual); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in Heavy Episodic Drinking | Through study completion, an average of monthly over 15 months
  Description Single Alcohol Screening Question (SASQ) (Williams and Vinson, 2001)
Change in Modal alcohol consumption | Through study completion, an average of monthly over 15 months
  Daily Drinking Questionnaire (DDQ) (Collins, Parks, & Marlatt, 1985)
Change in Negative Emotional State -- Depression | Through study completion, an average of monthly over 15 months
  The Patient Health Questionnaire (PHQ)-9

SECONDARY OUTCOMES:
Change in Alcohol-related problems | Through study completion, an average of monthly over 15 months
  Short Rutgers Alcohol Problems Index (S-RAPI) (Earleywine, LaBrie & Pedersen)
Change in Suicidal ideation | Through study completion, an average of monthly over 15 months
  Measure developed by Nock et al., 2007

OTHER OUTCOMES:
Change in Employment | Through study completion, an average of monthly over 15 months
  Current job situation/Change employment

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Bacharach, Ph.D., Principal Investigator — Cornell University
Locations (1):
- Joint Base Lewis-McChord, Tacoma, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Williams R, Vinson DC. Validation of a single screening question for problem drinking. J Fam Pract. 2001 Apr;50(4):307-12. PMID 11300981
- [Background] Collins RL, Parks GA, Marlatt GA. Social determinants of alcohol consumption: the effects of social interaction and model status on the self-administration of alcohol. J Consult Clin Psychol. 1985 Apr;53(2):189-200. doi: 10.1037//0022-006x.53.2.189. No abstract available. PMID 3998247
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Earleywine M, LaBrie JW, Pedersen ER. A brief Rutgers Alcohol Problem Index with less potential for bias. Addict Behav. 2008 Sep;33(9):1249-53. doi: 10.1016/j.addbeh.2008.05.006. Epub 2008 May 13. PMID 18547738
- [Background] Nock MK, Banaji MR. Prediction of suicide ideation and attempts among adolescents using a brief performance-based test. J Consult Clin Psychol. 2007 Oct;75(5):707-15. doi: 10.1037/0022-006X.75.5.707. PMID 17907852
- [Background] Morean ME, Kong G, Camenga DR, Cavallo DA, Connell C, Krishnan-Sarin S. First drink to first drunk: age of onset and delay to intoxication are associated with adolescent alcohol use and binge drinking. Alcohol Clin Exp Res. 2014 Oct;38(10):2615-21. doi: 10.1111/acer.12526. Epub 2014 Sep 24. PMID 25257574
- [Background] Saunders JB, Aasland OG, Babor TF, de la Fuente JR, Grant M. Development of the Alcohol Use Disorders Identification Test (AUDIT): WHO Collaborative Project on Early Detection of Persons with Harmful Alcohol Consumption--II. Addiction. 1993 Jun;88(6):791-804. doi: 10.1111/j.1360-0443.1993.tb02093.x. PMID 8329970
- [Background] Forbes D, Alkemade N, Mitchell D, Elhai JD, McHugh T, Bates G, Novaco RW, Bryant R, Lewis V. Utility of the Dimensions of Anger Reactions-5 (DAR-5) scale as a brief anger measure. Depress Anxiety. 2014 Feb;31(2):166-73. doi: 10.1002/da.22148. Epub 2013 Jun 25. PMID 23801571
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Britt TW, Adler AB, Sawhney G, Bliese PD. Coping Strategies as Moderators of the Association Between Combat Exposure and Posttraumatic Stress Disorder Symptoms. J Trauma Stress. 2017 Oct;30(5):491-501. doi: 10.1002/jts.22221. PMID 29078001
- [Background] Carver CS. You want to measure coping but your protocol's too long: consider the brief COPE. Int J Behav Med. 1997;4(1):92-100. doi: 10.1207/s15327558ijbm0401_6. PMID 16250744
- [Background] Sayer NA, Frazier P, Orazem RJ, Murdoch M, Gravely A, Carlson KF, Hintz S, Noorbaloochi S. Military to civilian questionnaire: a measure of postdeployment community reintegration difficulty among veterans using Department of Veterans Affairs medical care. J Trauma Stress. 2011 Dec;24(6):660-70. doi: 10.1002/jts.20706. Epub 2011 Dec 7. PMID 22162082
- [Background] Lindgren KP, Neighbors C, Teachman BA, Wiers RW, Westgate E, Greenwald AG. I drink therefore I am: validating alcohol-related implicit association tests. Psychol Addict Behav. 2013 Mar;27(1):1-13. doi: 10.1037/a0027640. Epub 2012 Mar 19. PMID 22428863
- [Background] Grant VV, Stewart SH, O'Connor RM, Blackwell E, Conrod PJ. Psychometric evaluation of the five-factor Modified Drinking Motives Questionnaire--Revised in undergraduates. Addict Behav. 2007 Nov;32(11):2611-32. doi: 10.1016/j.addbeh.2007.07.004. Epub 2007 Jul 13. PMID 17716823
- [Background] Ames GM, Grube JW. Alcohol availability and workplace drinking: mixed method analyses. J Stud Alcohol. 1999 May;60(3):383-93. doi: 10.15288/jsa.1999.60.383. PMID 10371267
- [Background] Ames GM, Grube JW, Moore RS. Social control and workplace drinking norms: a comparison of two organizational cultures. J Stud Alcohol. 2000 Mar;61(2):203-19. doi: 10.15288/jsa.2000.61.203. PMID 10757130
- [Background] Baer JS, Stacy A, Larimer M. Biases in the perception of drinking norms among college students. J Stud Alcohol. 1991 Nov;52(6):580-6. doi: 10.15288/jsa.1991.52.580. PMID 1758185
- [Background] Treloar H, Martens MP, McCarthy DM. The Protective Behavioral Strategies Scale-20: improved content validity of the Serious Harm Reduction subscale. Psychol Assess. 2015 Mar;27(1):340-6. doi: 10.1037/pas0000071. Epub 2015 Jan 5. PMID 25558969
- [Background] Nock MK, Wedig MM, Holmberg EB, Hooley JM. The emotion reactivity scale: development, evaluation, and relation to self-injurious thoughts and behaviors. Behav Ther. 2008 Jun;39(2):107-16. doi: 10.1016/j.beth.2007.05.005. Epub 2007 Oct 29. PMID 18502244
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] Bastien CH, Vallieres A, Morin CM. Validation of the Insomnia Severity Index as an outcome measure for insomnia research. Sleep Med. 2001 Jul;2(4):297-307. doi: 10.1016/s1389-9457(00)00065-4. PMID 11438246
- [Background] Hughes ME, Waite LJ, Hawkley LC, Cacioppo JT. A Short Scale for Measuring Loneliness in Large Surveys: Results From Two Population-Based Studies. Res Aging. 2004;26(6):655-672. doi: 10.1177/0164027504268574. PMID 18504506
- [Background] Brown DW, Balluz LS, Heath GW, Moriarty DG, Ford ES, Giles WH, Mokdad AH. Associations between recommended levels of physical activity and health-related quality of life. Findings from the 2001 Behavioral Risk Factor Surveillance System (BRFSS) survey. Prev Med. 2003 Nov;37(5):520-8. doi: 10.1016/s0091-7435(03)00179-8. PMID 14572437
- [Background] Bliese PD, Wright KM, Adler AB, Cabrera O, Castro CA, Hoge CW. Validating the primary care posttraumatic stress disorder screen and the posttraumatic stress disorder checklist with soldiers returning from combat. J Consult Clin Psychol. 2008 Apr;76(2):272-81. doi: 10.1037/0022-006X.76.2.272. PMID 18377123
- [Background] Rehm J, Greenfield TK, Walsh G, Xie X, Robson L, Single E. Assessment methods for alcohol consumption, prevalence of high risk drinking and harm: a sensitivity analysis. Int J Epidemiol. 1999 Apr;28(2):219-24. doi: 10.1093/ije/28.2.219. PMID 10342682
- [Background] Biener L, Abrams DB. The Contemplation Ladder: validation of a measure of readiness to consider smoking cessation. Health Psychol. 1991;10(5):360-5. doi: 10.1037//0278-6133.10.5.360. PMID 1935872
- [Background] Posner K, Brown GK, Stanley B, Brent DA, Yershova KV, Oquendo MA, Currier GW, Melvin GA, Greenhill L, Shen S, Mann JJ. The Columbia-Suicide Severity Rating Scale: initial validity and internal consistency findings from three multisite studies with adolescents and adults. Am J Psychiatry. 2011 Dec;168(12):1266-77. doi: 10.1176/appi.ajp.2011.10111704. PMID 22193671
- [Background] Nock MK, Holmberg EB, Photos VI, Michel BD. Self-Injurious Thoughts and Behaviors Interview: development, reliability, and validity in an adolescent sample. Psychol Assess. 2007 Sep;19(3):309-17. doi: 10.1037/1040-3590.19.3.309. PMID 17845122
- [Background] Nock MK, Hwang I, Sampson NA, Kessler RC. Mental disorders, comorbidity and suicidal behavior: results from the National Comorbidity Survey Replication. Mol Psychiatry. 2010 Aug;15(8):868-76. doi: 10.1038/mp.2009.29. Epub 2009 Mar 31. PMID 19337207
- [Background] Norman SB, Schmied E, Larson GE. Predictors of continued problem drinking and substance use following military discharge. J Stud Alcohol Drugs. 2014 Jul;75(4):557-66. doi: 10.15288/jsad.2014.75.557. PMID 24988254
- [Background] Conner KR, Bagge CL, Goldston DB, Ilgen MA. Alcohol and suicidal behavior: what is known and what can be done. Am J Prev Med. 2014 Sep;47(3 Suppl 2):S204-8. doi: 10.1016/j.amepre.2014.06.007. PMID 25145740
- [Background] Brenner LA, Barnes SM. Facilitating treatment engagement during high-risk transition periods: a potential suicide prevention strategy. Am J Public Health. 2012 Mar;102 Suppl 1(Suppl 1):S12-4. doi: 10.2105/AJPH.2011.300581. Epub 2012 Jan 25. No abstract available. PMID 22390585
- [Background] Kapur N, While D, Blatchley N, Bray I, Harrison K. Suicide after leaving the UK armed forces--a cohort study. PLoS Med. 2009 Mar 3;6(3):e26. doi: 10.1371/journal.pmed.1000026. PMID 19260757
- [Background] Cherpitel CJ, Borges GL, Wilcox HC. Acute alcohol use and suicidal behavior: a review of the literature. Alcohol Clin Exp Res. 2004 May;28(5 Suppl):18S-28S. doi: 10.1097/01.alc.0000127411.61634.14. PMID 15166633
- [Background] Schulenberg JE, Maggs JL. A developmental perspective on alcohol use and heavy drinking during adolescence and the transition to young adulthood. J Stud Alcohol Suppl. 2002 Mar;(14):54-70. doi: 10.15288/jsas.2002.s14.54. PMID 12022730
- [Background] Muthen BO, Muthen LK. The development of heavy drinking and alcohol-related problems from ages 18 to 37 in a U.S. national sample. J Stud Alcohol. 2000 Mar;61(2):290-300. doi: 10.15288/jsa.2000.61.290. PMID 10757140
- [Background] Karlamangla A, Zhou K, Reuben D, Greendale G, Moore A. Longitudinal trajectories of heavy drinking in adults in the United States of America. Addiction. 2006 Jan;101(1):91-9. doi: 10.1111/j.1360-0443.2005.01299.x. PMID 16393195
- [Background] Sher L, Braquehais MD, Casas M. Posttraumatic stress disorder, depression, and suicide in veterans. Cleve Clin J Med. 2012 Feb;79(2):92-7. doi: 10.3949/ccjm.79a.11069. PMID 22301558
- [Background] Thomas JL, Wilk JE, Riviere LA, McGurk D, Castro CA, Hoge CW. Prevalence of mental health problems and functional impairment among active component and National Guard soldiers 3 and 12 months following combat in Iraq. Arch Gen Psychiatry. 2010 Jun;67(6):614-23. doi: 10.1001/archgenpsychiatry.2010.54. PMID 20530011
- [Background] Finley EP, Bollinger M, Noel PH, Amuan ME, Copeland LA, Pugh JA, Dassori A, Palmer R, Bryan C, Pugh MJ. A national cohort study of the association between the polytrauma clinical triad and suicide-related behavior among US Veterans who served in Iraq and Afghanistan. Am J Public Health. 2015 Feb;105(2):380-7. doi: 10.2105/AJPH.2014.301957. PMID 25033126
- [Background] Cooper ML, Russell M, Skinner JB, Frone MR, Mudar P. Stress and alcohol use: moderating effects of gender, coping, and alcohol expectancies. J Abnorm Psychol. 1992 Feb;101(1):139-52. doi: 10.1037//0021-843x.101.1.139. PMID 1537960
- [Background] Carver CS, Scheier MF. Situational coping and coping dispositions in a stressful transaction. J Pers Soc Psychol. 1994 Jan;66(1):184-95. doi: 10.1037//0022-3514.66.1.184. PMID 8126648
- [Background] MacLean MG, Lecci L. A comparison of models of drinking motives in a university sample. Psychol Addict Behav. 2000 Mar;14(1):83-7. doi: 10.1037//0893-164x.14.1.83. PMID 10822750
- [Background] CONGER JJ. Alcoholism: theory, problem and challenge. II. Reinforcement theory and the dynamics of alcoholism. Q J Stud Alcohol. 1956 Jun;17(2):296-305. No abstract available. PMID 13336262
- [Background] Frone MR. Are work stressors related to employee substance use? The importance of temporal context assessments of alcohol and illicit drug use. J Appl Psychol. 2008 Jan;93(1):199-206. doi: 10.1037/0021-9010.93.1.199. PMID 18211145
- [Background] Hassija CM, Jakupcak M, Maguen S, Shipherd JC. The influence of combat and interpersonal trauma on PTSD, depression, and alcohol misuse in U.S. Gulf War and OEF/OIF women veterans. J Trauma Stress. 2012 Apr;25(2):216-9. doi: 10.1002/jts.21686. PMID 22522738
- [Background] Jones E, Fear NT. Alcohol use and misuse within the military: a review. Int Rev Psychiatry. 2011 Apr;23(2):166-72. doi: 10.3109/09540261.2010.550868. PMID 21521086
- [Background] Jacobson IG, Ryan MA, Hooper TI, Smith TC, Amoroso PJ, Boyko EJ, Gackstetter GD, Wells TS, Bell NS. Alcohol use and alcohol-related problems before and after military combat deployment. JAMA. 2008 Aug 13;300(6):663-75. doi: 10.1001/jama.300.6.663. PMID 18698065
- [Background] Sayer NA, Noorbaloochi S, Frazier P, Carlson K, Gravely A, Murdoch M. Reintegration problems and treatment interests among Iraq and Afghanistan combat veterans receiving VA medical care. Psychiatr Serv. 2010 Jun;61(6):589-97. doi: 10.1176/ps.2010.61.6.589. PMID 20513682
- [Background] Bandura A. Social learning of moral judgments. J Pers Soc Psychol. 1969 Mar;11(3):275-9. doi: 10.1037/h0026998. No abstract available. PMID 5784267
- [Background] Borsari B, Carey KB. Descriptive and injunctive norms in college drinking: a meta-analytic integration. J Stud Alcohol. 2003 May;64(3):331-41. doi: 10.15288/jsa.2003.64.331. PMID 12817821
- [Background] Larimer ME, Turner AP, Mallett KA, Geisner IM. Predicting drinking behavior and alcohol-related problems among fraternity and sorority members: examining the role of descriptive and injunctive norms. Psychol Addict Behav. 2004 Sep;18(3):203-12. doi: 10.1037/0893-164X.18.3.203. PMID 15482075
- [Background] Lewis MA, Litt DM, Blayney JA, Lostutter TW, Granato H, Kilmer JR, Lee CM. They drink how much and where? Normative perceptions by drinking contexts and their association to college students' alcohol consumption. J Stud Alcohol Drugs. 2011 Sep;72(5):844-53. doi: 10.15288/jsad.2011.72.844. PMID 21906511
- [Background] Frone MR. Predictors of overall and on-the-job substance use among young workers. J Occup Health Psychol. 2003 Jan;8(1):39-54. doi: 10.1037//1076-8998.8.1.39. PMID 12553528
- [Background] Hammen C. Stress and depression. Annu Rev Clin Psychol. 2005;1:293-319. doi: 10.1146/annurev.clinpsy.1.102803.143938. PMID 17716090
- [Background] McGonagle KA, Kessler RC. Chronic stress, acute stress, and depressive symptoms. Am J Community Psychol. 1990 Oct;18(5):681-706. doi: 10.1007/BF00931237. PMID 2075897
- [Background] Toker S, Biron M. Job burnout and depression: unraveling their temporal relationship and considering the role of physical activity. J Appl Psychol. 2012 May;97(3):699-710. doi: 10.1037/a0026914. Epub 2012 Jan 9. PMID 22229693
- [Background] Brown GP, Hammen CL, Craske MG, Wickens TD. Dimensions of dysfunctional attitudes as vulnerabilities to depressive symptoms. J Abnorm Psychol. 1995 Aug;104(3):431-5. doi: 10.1037//0021-843x.104.3.431. PMID 7673566
- [Background] Finlay-Jones R, Brown GW. types of stressful life event and the onset of anxiety and depressive disorders. Psychol Med. 1981 Nov;11(4):803-15. doi: 10.1017/s0033291700041301. PMID 7323236
- [Background] Hobfoll SE. Conservation of resources. A new attempt at conceptualizing stress. Am Psychol. 1989 Mar;44(3):513-24. doi: 10.1037//0003-066x.44.3.513. PMID 2648906
- [Background] Hobfoll SE, Johnson RJ, Ennis N, Jackson AP. Resource loss, resource gain, and emotional outcomes among inner city women. J Pers Soc Psychol. 2003 Mar;84(3):632-43. PMID 12635922
- [Background] Holahan CJ, Moos RH, Holahan CK, Cronkite RC. Resource loss, resource gain, and depressive symptoms: a 10-year model. J Pers Soc Psychol. 1999 Sep;77(3):620-9. doi: 10.1037//0022-3514.77.3.620. PMID 10510511
- [Background] Kaniasty K, Norris FH. A test of the social support deterioration model in the context of natural disaster. J Pers Soc Psychol. 1993 Mar;64(3):395-408. doi: 10.1037//0022-3514.64.3.395. PMID 8468668
- [Background] Stout RL, Wirtz PW, Carbonari JP, Del Boca FK. Ensuring balanced distribution of prognostic factors in treatment outcome research. J Stud Alcohol Suppl. 1994 Dec;12:70-5. doi: 10.15288/jsas.1994.s12.70. PMID 7723001
- [Background] Cosper R. Drinking as conformity; a critique of sociological literature on occupational differences in drinking. J Stud Alcohol. 1979 Sep;40(9):868-91. doi: 10.15288/jsa.1979.40.868. PMID 513778
- [Background] Guttmannova K, Hill KG, Bailey JA, Lee JO, Hartigan LA, Hawkins JD, Catalano RF. Examining explanatory mechanisms of the effects of early alcohol use on young adult alcohol dependence. J Stud Alcohol Drugs. 2012 May;73(3):379-90. doi: 10.15288/jsad.2012.73.379. PMID 22456243
- [Background] Neighbors C, Lewis MA, Atkins DC, Jensen MM, Walter T, Fossos N, Lee CM, Larimer ME. Efficacy of web-based personalized normative feedback: a two-year randomized controlled trial. J Consult Clin Psychol. 2010 Dec;78(6):898-911. doi: 10.1037/a0020766. PMID 20873892
- [Background] Neighbors C, Larimer ME, Lewis MA. Targeting misperceptions of descriptive drinking norms: efficacy of a computer-delivered personalized normative feedback intervention. J Consult Clin Psychol. 2004 Jun;72(3):434-47. doi: 10.1037/0022-006X.72.3.434. PMID 15279527
- [Background] Lewis MA, Neighbors C, Oster-Aaland L, Kirkeby BS, Larimer ME. Indicated prevention for incoming freshmen: personalized normative feedback and high-risk drinking. Addict Behav. 2007 Nov;32(11):2495-508. doi: 10.1016/j.addbeh.2007.06.019. Epub 2007 Jun 28. PMID 17658695
- [Background] Lewis MA, Neighbors C. Optimizing personalized normative feedback: the use of gender-specific referents. J Stud Alcohol Drugs. 2007 Mar;68(2):228-37. doi: 10.15288/jsad.2007.68.228. PMID 17286341
- [Background] Geisner IM, Neighbors C, Larimer ME. A randomized clinical trial of a brief, mailed intervention for symptoms of depression. J Consult Clin Psychol. 2006 Apr;74(2):393-9. doi: 10.1037/0022-006X.74.2.393. PMID 16649884
- [Background] Geisner IM, Koopmann J, Bamberger P, Wang M, Larimer ME, Nahum-Shani I, Bacharach S. When the party continues: Impulsivity and the effect of employment on young adults' post-college alcohol use. Addict Behav. 2018 Feb;77:114-120. doi: 10.1016/j.addbeh.2017.09.014. Epub 2017 Sep 28. PMID 28992576
- [Background] Saunders JB, Kypri K, Walters ST, Laforge RG, Larimer ME. Approaches to brief intervention for hazardous drinking in young people. Alcohol Clin Exp Res. 2004 Feb;28(2):322-9. doi: 10.1097/01.alc.0000113418.12889.08. PMID 15112940